CLINICAL TRIAL: NCT01450306
Title: Exposure, D-cycloserine Enhancement, and Functional Magnetic Resonance Imaging (fMRI) in Snake Phobics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hartford Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NAVE003220HU
Record Dates: First submitted 2011-10-06; First posted 2011-10-12 (Estimated); Results first posted 2016-04-21 (Estimated); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Specific Phobia
MeSH Terms: conditions — Phobia, Specific | interventions — Cycloserine; Implosive Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- D-cycloserine plus exposure therapy (Experimental): Single session (up to 3 hr) of in vivo exposure therapy plus 50 mg oral d-cycloserine administered 1 hr prior to exposure therapy session
  Interventions: Drug: D-cycloserine; Behavioral: Exposure therapy
- Placebo plus exposure therapy (Placebo Comparator): Single session (up to 3 hr) of in vivo exposure therapy plus oral placebo capsule administered 1 hr prior to exposure therapy session
  Interventions: Behavioral: Exposure therapy; Drug: Placebo

INTERVENTIONS:
Drug: D-cycloserine — 50 mg d-cycloserine, oral, 1 dose
  Arms: D-cycloserine plus exposure therapy
Behavioral: Exposure therapy — Single session graded in vivo exposure therapy, 60-180 minutes
Drug: Placebo — Single capsule of oral placebo, administered once 1 hr prior to exposure therapy
  Arms: Placebo plus exposure therapy

SUMMARY:
The aim of the present study is to determine whether people receiving d-cycloserine and exposure therapy show different brain reactions to symptom provocation compared to people receiving placebo and exposure therapy.

DETAILED DESCRIPTION:
D-cycloserine (DCS) is a partial N-methyl-D-aspartate (NMDA) receptor agonist that may improve or accelerate extinction learning. We will randomly assign people with snake phobia to receive DCS or placebo, and then provide all participants with exposure therapy. We will examine whether people receiving DCS and vs. placebo show different brain reactions to symptom provocation before and after exposure therapy.

ELIGIBILITY:
Inclusion Criteria:

* Primary diagnosis of specific phobia (snakes)

Exclusion Criteria:

* History of psychosis, obsessive-compulsive disorder, or mania
* Recent substance abuse or suicidality
* Previous receipt of study treatments

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-07; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Tolin, PhD, Principal Investigator — Hartford Hospital
Locations (1):
- Institute of Living/Hartford Hospital, Hartford, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be made available upon request

REFERENCES:
- [Result] Nave AM, Tolin DF, Stevens MC. Exposure therapy, D-cycloserine, and functional magnetic resonance imaging in patients with snake phobia: a randomized pilot study. J Clin Psychiatry. 2012 Sep;73(9):1179-86. doi: 10.4088/JCP.11m07564. PMID 23059145

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | D-cycloserine Plus Exposure Therapy | Placebo Plus Exposure Therapy
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | D-cycloserine Plus Exposure Therapy | Placebo Plus Exposure Therapy | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 10 | 20
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 39 (13.91) | 34.6 (12.69) | 37 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 12
  Male | 4 | 4 | 8
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Snake Questionnaire (SNAQ)
Description: 30-item self-report scale of severity of snake fear and avoidance
  Range: 0-30; higher values indicate greater fear severity
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | D-cycloserine Plus Exposure Therapy | Placebo Plus Exposure Therapy
Number analyzed (Participants) | 10 | 10
units on a scale | 9.6 (5.99) | 9.7 (6.18)

2. Secondary Outcome: Clinician's Global Impression (CGI)-Severity
Description: Clinician rating of global illness severity (at pre- and post-treatment)
  CGI-Severity range 1-7; higher scores indicate greater illness severity.
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | D-cycloserine Plus Exposure Therapy | Placebo Plus Exposure Therapy
Number analyzed (Participants) | 10 | 10
units on a scale | 3 (1.15) | 2.7 (.68)

3. Secondary Outcome: Clinician's Global Impression (CGI)-Improvement
Description: Clinician rating of global illness severity (at post-treatment)
  CGI-Improvement range 1-7; higher scores indicate poorer improvement; classified as responder if score = 1 or 2, nonresponder if score > 2
Time Frame: 2 weeks
Measure: Number; unit: participants
Arm/Group | D-cycloserine Plus Exposure Therapy | Placebo Plus Exposure Therapy
Number analyzed (Participants) | 10 | 10
participants | 8 | 9

ADVERSE EVENTS:
Arm/Group | D-cycloserine Plus Exposure Therapy | Placebo Plus Exposure Therapy
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 1/10 | 0/10
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | D-cycloserine Plus Exposure Therapy (N=10) | Placebo Plus Exposure Therapy (N=10)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) — Mild nausea, resolved without intervention

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes